CLINICAL TRIAL: NCT00136435
Title: A Multicenter Phase II Study in Adults With Untreated Acute Lymphoblastic Leukemia: Testing Pharmacokinetically Individualized Doses of L-Asparaginase Following the Dana Farber Cancer Institute (DFCI) Pediatric Consortium Protocol
Brief Title: A Study in Adults With Untreated Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Daniel J. DeAngelo, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-175
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; acute lymphoblastic leukemia; chemotherapy; asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisone; Doxorubicin; Vincristine; Methotrexate; Asparaginase; Dexamethasone; Leucovorin; Cytarabine; Hydrocortisone; Mercaptopurine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Only Arm for this study (Other): Only Arm for this study
  Interventions: Drug: prednisone; Drug: doxorubicin; Drug: vincristine; Drug: methotrexate; Drug: asparaginase; Drug: dexamethasone; Radiation: cranial radiation; Drug: leucovorin; Drug: cytarabine; Drug: hydrocortisone; Drug: 6-mercaptopurine (6-MP); Drug: e. coli L-asparaginase

INTERVENTIONS:
Drug: prednisone — Induction Phase: Given orally on days 1-28
Drug: doxorubicin — Induction Phase: Given intravenously on day 1 and day 2 CNS Therapy: Given intravenously on day 1 Intensification: Given day 1 of each cycle
Drug: vincristine — Induction: Given intravenously on days 1, 8, 15, and 22. If complete remission not achieved, will be given on days 29, 36 and 43.
  CNS Therapy: Given intravenously on day 1. Intensification: Given intravenously on day 1 of each cycle. Continuation: Given intravenously on day 1 of each cycle
Drug: methotrexate — Induction: Given intravenously on day 3. CNS Therapy: Given intrathecally 4 times over two weeks Intensification: Given intrathecally every 18 weeks Continuation: Given intravenously weekly and intrathecally every 18 weeks
Drug: asparaginase — Induction: Given into the muscle on day 5
Drug: dexamethasone — Intensification: Given orally on days 1-5 of each cycle
Radiation: cranial radiation — Given in 10 daily treatments during CNS therapy phase
Drug: leucovorin — Induction: Given intravenously or orally 36 hours after methotrexate
Drug: cytarabine — Induction: Given intrathecally days 1, 15, 29 CNS Therapy: Given intrathecally 4 times over 2 weeks Intensification: Given intrathecally every 18 weeks Continuation: Given intrathecally every 18 weeks
  Other Names: Ara-C
Drug: hydrocortisone — Induction: Given intrathecally on days 15 and 29. Intensification: Given intrathecally every 18 weeks. Continuation: Given intrathecally every 18 weeks.
Drug: 6-mercaptopurine (6-MP) — CNS Therapy: Taken orally on days 1-14. Intensification: Taken orally on days 1-14. Continuation: Taken orally on days 1-14.
Drug: e. coli L-asparaginase — Intensification: Given in to the muscle weekly.

SUMMARY:
The purpose of this study is to determine the safety and optimal dosing of L-asparaginase in adult patients with acute lymphoblastic leukemia (ALL) between the ages of 18 and 50 years.

DETAILED DESCRIPTION:
This study has four treatment phases: 1) induction, 2) central nervous system therapy, 3) intensification, and 4) continuation.

The induction phase lasts one month and eight drugs are used during this phase of treatment. The drugs are administered as follows:

* Prednisone; on days 1-28:
* Vincristine; on days 1, 8, 15, and 22:
* Doxorubicin; on days 1 and 2:
* Methotrexate; on day 3;
* Leucovorin; 36 hours after methotrexate:
* Asparaginase; on day 5:
* Intra-thecal Cytarabine; on days 1, 15, and 29:
* Intra-thecal Methotrexate/Hydrocortisone; on days 15 and 29

A bone marrow aspirate and biopsy will be obtained on day 15 and day 29 of induction therapy. If on day 29, the patients' bone marrow and peripheral blood counts are not in complete remission, then the patient may receive vincristine on days 29, 36 and 43. Bone marrow biopsy will be repeated weekly until complete remission is documented. If the patient does not achieve complete remission by day 49, they will be removed from the study.

Central nervous system (CNS) therapy begins immediately after the end of the induction therapy. This phase of treatment should last 3 weeks. Treatment includes a series of spinal taps with the instillation of anti-leukemia drugs. Four spinal taps will be performed over a two week period. Anti-leukemia drugs will also be given orally. The drugs given are as follows: Vincristine; on day 1: Doxorubicin; on day 1: 6-mercaptopurine (6-MP); on days 1-14: Intra-thecal Methotrexate/Cytarabine; 4 times over 2 weeks.

Radiation therapy (RT) will be delivered in 10 daily treatments during the CNS phase of therapy.

The intensification phase begins as soon as the CNS phase ends and lasts approximately 30 weeks. It consists of cycles of chemotherapy repeated every 3 weeks, along with asparaginase administered weekly. The drugs given are as follows: Vincristine; day 1: Dexamethasone; days 1-5: 6-MP; days 1-14: Doxorubicin; day 1: Asparaginase; weekly: Methotrexate; weekly: Intra-thecal Hydrocortisone/Methotrexate/cytarabine; every 18 weeks.

The continuation phase of treatment begins after the intensification phase. It consists of cycles of chemotherapy repeated every three weeks and will last until the patient is in remission for two years. The drugs given are: Vincristine; day 1 : Prednisone or Dexamethasone; days 1-5: 6-MP; days 1-14: Methotrexate; weekly: Intra-thecal Methotrexate/Cytarabine/Hydrocortisone: every 18 weeks.

During this study, blood tests will be performed at the start of therapy, at day 29 post induction and at the time of each intra-thecal therapy (every 18 weeks).

Bone marrow biopsy/aspirate will be done days 15 and 29 of induction, then every 6 months until completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically documented acute lymphoblastic leukemia, excluding mature B-cell ALL.
* No prior therapy for leukemia with the following exceptions:

  * up to one week of steroids;
  * emergent leukapheresis;
  * emergency treatment for hyperleukocytosis with hydroxyurea;
  * cranial RT for CNS leukostasis (one dose only);
  * emergent radiation therapy to the mediastinum.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Between the ages of 18 to 50 years.

Exclusion Criteria:

* Uncontrolled active infection.
* Pregnancy or nursing mothers.
* Prior history of pancreatitis.
* Prior history of a cerebrovascular accident or hemorrhage.
* Evidence of infection with the human immunodeficiency virus.
* Active psychiatric or mental illness making informed consent or careful clinical follow-up unlikely.
* The treating physician should consider all relevant medical and other considerations when deciding whether this protocol is appropriate for a particular patient.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2002-06; Primary Completion 2008-11 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. DeAngelo, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Of Columbia Medical Center, New York, New York
- Canada (9):
  - Manitoba Blood & Marrow Transplant Program CancerCare Manitoba, Winnipeg, Manitoba
  - McMaster University Medical Center, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Queen Elizabeth II, Halifax

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase: prednisone: Induction Phase: Orally days 1-28
  doxorubicin: Induction Phase: Intravenously days 1 and 2 CNS Therapy: Intravenously day 1 Intensification: Given day 1 of each cycle
  vincristine: Induction: Intravenously days 1, 8, 15, and 22. If complete remission not achieved, will be given on days 29, 36 and 43.
  CNS Therapy: Intravenously day 1. Intensification: Intravenously day 1 of each cycle. Continuation: Intravenously day 1 of each cycle
  methotrexate: Induction: Intravenously day 3. CNS Therapy: Intrathecally 4x over two weeks Intensification: Intrathecally every 18 weeks Continuation: Intravenously weekly and intrathecally every 18 weeks
  asparaginase: Induction: Given into the muscle on day 5
  dexamethasone: Intensification: Orally days 1-5 of each cycle
  cranial radiation: 10 daily treatments during CNS phase
  leucovorin: Induction: Intravenously/orally 36 hours after methotrexate
  cytarabine: Induction: Intrathecally days 1, 15, 29 CNS Therapy: Intrathecally 4x over 2 weeks Intensification: Intrathecally every 18 weeks Continuation: Intrathecally every 18 weeks
  hydrocortisone: Induction: Intrathecally days 15 and 29. Intensification: Intrathecally every 18 weeks. Continuation: Intrathecally every 18 weeks.
  6-mercaptopurine (6-MP): CNS Therapy: Orally days 1-14. Intensification: Orally on days 1-14. Continuation: Orally on days 1-14.
  e. coli L-asparaginase: Intensification: Given in to the muscle weekly.
Period: Overall Study
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Started | 100
Started Study Treatment (2 patients were removed from study prior to receiving any chemotherapy, as they were found to have bilineage leukemia.) | 98
Eligible and Treated | 92
Achieved Complete Remission | 78
Initiated Asparaginase Consolidation Therapy | 57
Completed | 36
Not Completed | 64
Not completed — Ineligible | 8
Not completed — Induction Death | 1
Not completed — Induction Failure | 10
Not completed — Withdrew prior to initiating imatinib/Ph+ | 3
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 19
Not completed — Relapse | 4
Not completed — Transplant in first Complete Remission (CR) | 16

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Number analyzed (Participants) | 100
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 49
  30-50 years | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 88
  More than one race | 0
  Unknown or Not Reported | 5
Immunophenotype [Count of Participants; unit: Participants]
  B-cell | 81
  T-cell | 19
White Blood Count (WBC) (x 10^-3) at diagnosis [Count of Participants; unit: Participants]
  < 20 | 60
  >/= 20 | 39
  Unknown | 1
Central Nervous System (CNS) status at diagnosis [Count of Participants; unit: Participants]
  CNS 1 (-) CSF WBC <5 without blasts | 83
  CNS 2 (+) CSF WBC <5 with blasts | 6
  CNS 3 (+) CSF WBC >=5 with blasts | 1
  Unknown | 10
Eastern Cooperative Oncology Group (ECOG) Risk classification [Count of Participants; unit: Participants] — ECOG risk is defined as follows: HR includes any patients with an MLL rearrangement or Ph+ and B-cell patients with WBC ≥ 35K or age ≥ 35 years and T-cell patients with WBC ≥ 100K.
  Participants
    Standard Risk (SR) | 42
    High Risk (HR) | 58

OUTCOME MEASURES:

1. Primary Outcome: Asparaginase Completion Rate
Description: Feasibility based on the rate of asparaginase completion defined as the percentage of patients who, after having achieved a complete remission after induction therapy, complete all 30 doses of asparaginase as part of intensification therapy. Complete remission is defined as peripheral blood without lymphoblasts, a bone marrow with <5% lymphoblasts, an antigen-presenting cell (APC) > 1000/mm3, platelets > 100,000/mm3, and no evidence of extramedullary leukemia.
Time Frame: Assessed at the end of the 30-week post-induction treatment period or when the participant comes off treatment, whichever occurs first.
Population: The analysis dataset is comprised of all patients who initiated asparaginase consolidation therapy.
Measure: Number (80% Confidence Interval); unit: Percentage of patients
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Number analyzed (Participants) | 57
Percentage of patients | 63 [54 to 72]

2. Secondary Outcome: 4-year Disease-Free Survival
Description: Disease-Free Survival (DFS) based on the Kaplan-Meier method is defined as the time from achieving a complete remission to the first of disease recurrence or death, censored at time of last disease assessment. 4-year DFS is the percent probability of patients remaining alive, relapse-free and without occurrence of second malignant neoplasm 4 years from complete remission. Disease relapse is defined as >25% lymphoblasts identified morphologically in bone marrow aspirate/biopsy, or identification of lymphoblasts in marrow (any percentage) identified to be leukemic by flow cytometry, cytogenetics, fluorescent in situ hybridization (FISH), immunohistochemistry, or other tests. Appearance of leukemic cells at any extramedullary site (a single, unequivocal lymphoblast in the cerebrospinal fluid (CSF) may qualify as CNS leukemia) also qualifies if confirmed by the PI.
Time Frame: Assessed continuously throughout the treatment period, and annually for 5 years following the completion of protocol treatment, (up to 5 years). Relevant for this measure is 4 years from the date of complete remission.
Population: The analysis dataset is comprised of all eligible patients who achieved a CR.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Number analyzed (Participants) | 78
Percent probability | 69 [56 to 78]

3. Secondary Outcome: 4-year Overall Survival
Description: Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death from any cause, and will be censored the date last known alive. 4-year OS is the percent probability of patients remaining alive 4 years from study entry.
Time Frame: Assessed continuously throughout the treatment period, and annually for 5 years following the completion of protocol treatment (unless the participant dies or is lost to follow-up). Median follow-up for the whole trial is 4.5 years (95% CI:4.1-5.0 years).
Population: The analysis dataset is comprised of all eligible patients.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Number analyzed (Participants) | 92
Percent probability | 67 [56 to 76]

4. Secondary Outcome: 4-year Event-Free Survival
Description: Event-Free Survival (EFS) based on the Kaplan-Meier method is defined as the time from study entry to the first event of death during induction therapy, failure to achieve CR at the end of induction, death during remission, or relapse. 4-year EFS is the percent probability of patients remaining alive, relapse-free and without occurrence of second malignant neoplasm 4 years from study entry. Patients not achieving a CR will be considered events at time zero. EFS will be censored at time of last disease assessment. Disease relapse is defined as >25% lymphoblasts identified morphologically in bone marrow aspirate/biopsy, or identification of lymphoblasts in marrow (any percentage) identified to be leukemic by flow cytometry, cytogenetics, FISH, immunohistochemistry, or other tests. Appearance of leukemic cells at any extramedullary site (a single, unequivocal lymphoblast in the CSF may qualify as CNS leukemia) also qualifies if confirmed by the PI.
Time Frame: as for outcome 3
Population: The analysis dataset is comprised of all eligible patients.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Number analyzed (Participants) | 92
Percent probability | 58 [47 to 68]

5. Secondary Outcome: Post-Induction Nadir Serum Asparaginase Activity Level
Description: Nadir serum asparaginase activity (NSAA) levels were estimated based on established methods.
Time Frame: Samples for nadir serum asparaginase activity levels were assayed prior to asparaginase dose given during post-induction, at Weeks 2, 4, 7, 10, 13, 16, 19, 22, 25, 28, and 30.
Population: The analysis dataset is comprised of all eligible patients for whom serum asparaginase activity levels were assayed.
Measure: Median (Full Range); unit: IU/ml
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Number analyzed (Participants) | 92
IU/ml
  Week 2 NSAA Level: number analyzed (Participants) | 43
  Week 2 NSAA Level | 0 [0.0 to 0.172]
  Week 4 NSAA Level: number analyzed (Participants) | 39
  Week 4 NSAA Level | 0.047 [0.0 to 0.318]
  Week 7 NSAA Level: number analyzed (Participants) | 34
  Week 7 NSAA Level | 0.0825 [0.0 to 0.661]
  Week 10 NSAA Level: number analyzed (Participants) | 37
  Week 10 NSAA Level | 0.088 [0.0 to 0.353]
  Week 13 NSAA Level: number analyzed (Participants) | 30
  Week 13 NSAA Level | 0.118 [0.0 to 0.315]
  Week 16 NSAA Level: number analyzed (Participants) | 31
  Week 16 NSAA Level | 0.069 [0.0 to 0.259]
  Week 19 NSAA Level: number analyzed (Participants) | 28
  Week 19 NSAA Level | 0.075 [0.0 to 0.248]
  Week 22 NSAA Level: number analyzed (Participants) | 28
  Week 22 NSAA Level | 0.0865 [0.0 to 0.443]
  Week 25 NSAA Level: number analyzed (Participants) | 30
  Week 25 NSAA Level | 0.0925 [0.0 to 0.236]
  Week 28 NSAA Level: number analyzed (Participants) | 24
  Week 28 NSAA Level | 0.072 [0.0 to 0.255]
  Week 30 NSAA Level: number analyzed (Participants) | 21
  Week 30 NSAA Level | 0.065 [0.0 to 0.249]

6. Secondary Outcome: Number of Participants With Asparaginase-Related Toxicity
Description: Asparaginase-related toxicity rate is defined as the percentage of patients who experience allergy (all grades), pancreatitis, thrombotic or bleeding complications, bone fracture, or avascular necrosis based on Common Terminology Criteria for Adverse Events (CTCAE) v2.
Time Frame: Assessed on an ongoing basis (at least once every 3 months) while patient is on study, and including the treatment phases of Induction, CNS, Intensification, and Continuation. Treatment duration for this study was a median (range) of 507 days (0-1097).
Population: The analysis dataset is comprised of all eligible patients.
Measure: Number; unit: participants
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
Number analyzed (Participants) | 92
participants
  Overall Number of Participants with Pancreatitis | 10
  Overall Number of Participants with Allergy/rash | 5
  Overall Number of Participants with Thrombosis/embolism | 16
  Overall Number of Participants with Bone fracture | 7
  Overall Number of Participants with Avascular necrosis | 5
  Number of Participants with Pancreatitis in Induction | 1
  Number of Participants with Allergy/rash in Induction | 1
  Number of Participants with Thrombosis/embolism in Induction | 1
  Number of Participants with Bone fracture in Induction | 0
  Number of Participants with Avascular necrosis in Induction | 0
  Number of Participants with Pancreatitis in Intensification: number analyzed (Participants) | 62
  Number of Participants with Pancreatitis in Intensification | 8
  Number of Participants with Allergy/rash in Intensification: number analyzed (Participants) | 62
  Number of Participants with Allergy/rash in Intensification | 4
  Number of Participants with Thrombosis/embolism in Intensification: number analyzed (Participants) | 62
  Number of Participants with Thrombosis/embolism in Intensification | 14
  Number of Participants with Bone fracture in Intensification: number analyzed (Participants) | 62
  Number of Participants with Bone fracture in Intensification | 3
  Number of Participants with Avascular necrosis in Intensification: number analyzed (Participants) | 62
  Number of Participants with Avascular necrosis in Intensification | 2
  Number of Participants with Pancreatitis in Continuation: number analyzed (Participants) | 48
  Number of Participants with Pancreatitis in Continuation | 2
  Number of Participants with Allergy/rash in Continuation: number analyzed (Participants) | 48
  Number of Participants with Allergy/rash in Continuation | 0
  Number of Participants with Thrombosis/embolism in Continuation: number analyzed (Participants) | 48
  Number of Participants with Thrombosis/embolism in Continuation | 2
  Number of Participants with Bone fracture in Continuation: number analyzed (Participants) | 48
  Number of Participants with Bone fracture in Continuation | 5
  Number of Participants with Avascular necrosis in Continuation: number analyzed (Participants) | 48
  Number of Participants with Avascular necrosis in Continuation | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were continuously monitored and reported every 3 months during treatment. Adverse events were monitored for the treatment duration of this study, which was a median (range) of 507 days (0-1097). All-Cause Mortality was monitored for the duration of follow-up for this study, which was a median (range) of 3.2 (0-7.9) years. Data is reported for the entire study cohort.
Description: Reporting included all observed adverse events, with grade and attribution to study treatment. Maximum grade by type was calculated with serious adverse events defined as either 1) G5, 2) G4 unless myelosuppression or unequivocally due to disease or considered expected for chemotherapy drugs used, 3) G2 or G3 events that are unexpected and Possibly, Probably, or Definitely related to study treatment. Since SAE data was not collected separately, all AEs have been reported in the SAE table.
Arm/Group | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase
All-Cause Mortality (participants affected / at risk) | 40/98
Serious Adverse Events (participants affected / at risk) | 98/98
Other Adverse Events (participants affected / at risk) | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction, CNS, and Intensification With Pharmacokinetically Individualized Doses of L-asparaginase (N=98)
Anemia (Blood and lymphatic system disorders) | 94
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 18
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 30
Cardiac disorders - Other, specify (Cardiac disorders) | 56
Palpitations (Cardiac disorders) | 4
Sinus bradycardia (Cardiac disorders) | 5
Sinus tachycardia (Cardiac disorders) | 22
Ventricular arrhythmia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 8
Ear pain (Ear and labyrinth disorders) | 9
Hearing impaired (Ear and labyrinth disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Cushingoid (Endocrine disorders) | 22
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 11
Cataract (Eye disorders) | 8
Conjunctivitis (Eye disorders) | 5
Dry eye (Eye disorders) | 1
Extraocular muscle paresis (Eye disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 10
Glaucoma (Eye disorders) | 1
Night blindness (Eye disorders) | 1
Photophobia (Eye disorders) | 4
Watering eyes (Eye disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 55
Ascites (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 51
Diarrhea (Gastrointestinal disorders) | 65
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 32
Dysphagia (Gastrointestinal disorders) | 35
Dysphasia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 10
Gastric hemorrhage (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 41
Ileus (Gastrointestinal disorders) | 4
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 71
Nausea (Gastrointestinal disorders) | 83
Pancreatitis (Gastrointestinal disorders) | 11
Proctitis (Gastrointestinal disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 20
Rectal pain (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 76
Chills (General disorders) | 24
Fatigue (General disorders) | 82
Fever (General disorders) | 27
General disorders and administration site conditions - Other, specify (General disorders) | 15
Injection site reaction (General disorders) | 9
Non-cardiac chest pain (General disorders) | 19
Pain (General disorders) | 66
Hepatic failure (Hepatobiliary disorders) | 3
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 10
Anaphylaxis (Immune system disorders) | 6
Immune system disorders - Other, specify (Immune system disorders) | 8
Catheter related infection (Infections and infestations) | 8
Infections and infestations - Other, specify (Infections and infestations) | 74
Wound infection (Infections and infestations) | 7
Bruising (Injury, poisoning and procedural complications) | 15
Dermatitis radiation (Injury, poisoning and procedural complications) | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 7
Activated partial thromboplastin time prolonged (Investigations) | 18
Alanine aminotransferase increased (Investigations) | 90
Alkaline phosphatase increased (Investigations) | 19
Aspartate aminotransferase increased (Investigations) | 89
Blood bilirubin increased (Investigations) | 72
CPK increased (Investigations) | 2
Cardiac troponin I increased (Investigations) | 2
Cardiac troponin T increased (Investigations) | 1
Cholesterol high (Investigations) | 16
Creatinine increased (Investigations) | 30
Fibrinogen decreased (Investigations) | 74
GGT increased (Investigations) | 3
INR increased (Investigations) | 16
Investigations - Other, specify (Investigations) | 17
Lipase increased (Investigations) | 8
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 94
Platelet count decreased (Investigations) | 91
Serum amylase increased (Investigations) | 9
Weight gain (Investigations) | 4
Weight loss (Investigations) | 17
White blood cell decreased (Investigations) | 23
Acidosis (Metabolism and nutrition disorders) | 6
Alkalosis (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 70
Dehydration (Metabolism and nutrition disorders) | 20
Hypercalcemia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 83
Hyperkalemia (Metabolism and nutrition disorders) | 14
Hypermagnesemia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 17
Hypertriglyceridemia (Metabolism and nutrition disorders) | 19
Hyperuricemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 30
Hypocalcemia (Metabolism and nutrition disorders) | 27
Hypoglycemia (Metabolism and nutrition disorders) | 17
Hypokalemia (Metabolism and nutrition disorders) | 21
Hypomagnesemia (Metabolism and nutrition disorders) | 26
Hyponatremia (Metabolism and nutrition disorders) | 25
Hypophosphatemia (Metabolism and nutrition disorders) | 21
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 35
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 30
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 26
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 36
Myalgia (Musculoskeletal and connective tissue disorders) | 49
Myositis (Musculoskeletal and connective tissue disorders) | 2
Arachnoiditis (Nervous system disorders) | 3
Ataxia (Nervous system disorders) | 14
Cognitive disturbance (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 48
Dysgeusia (Nervous system disorders) | 19
Extrapyramidal disorder (Nervous system disorders) | 2
Headache (Nervous system disorders) | 75
Intracranial hemorrhage (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 22
Neuralgia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 16
Peripheral sensory neuropathy (Nervous system disorders) | 66
Seizure (Nervous system disorders) | 8
Syncope (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 8
Vasovagal reaction (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 37
Confusion (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 42
Euphoria (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 55
Personality change (Psychiatric disorders) | 2
Psychosis (Psychiatric disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 4
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 10
Urinary frequency (Renal and urinary disorders) | 11
Urinary incontinence (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 4
Urinary tract pain (Renal and urinary disorders) | 7
Urine discoloration (Renal and urinary disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 3
Irregular menstruation (Reproductive system and breast disorders) | 3
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 3
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 5
Vaginal inflammation (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 17
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 52
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 36
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 54
Dry skin (Skin and subcutaneous tissue disorders) | 12
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 30
Nail loss (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Purpura (Skin and subcutaneous tissue disorders) | 26
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 47
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 48
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 4
Flushing (Vascular disorders) | 7
Hot flashes (Vascular disorders) | 8
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 17
Phlebitis (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 25
Vascular disorders - Other, specify (Vascular disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes